CLINICAL TRIAL: NCT01008683
Title: Antibody Production Following H1N1 Influenza Vaccination After Stem Cell and Heart Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Dan Engelhard, HMO
Other Study IDs: engelhard-HMO-CTIL
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2009-11-06 (Estimated); Status verified 2009-11

CONDITIONS: H1N1 Influenza
Keywords: Stem cell and and heart transplant patients who will receive pandemic H1N1 influenza vaccinations
MeSH Terms: conditions — Orthomyxoviridae Infections

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stem cell and and heart transplant patients: Stem cell and and heart transplant patients

SUMMARY:
Stem cell and and heart transplant patients will receive pandemic H1N1 influenza vaccination according to the clinical guidelines.

In these patients the investigators will measure the specific antibody production.

DETAILED DESCRIPTION:
Stem cell and and heart transplant patients will receive pandemic H1N1 influenza vaccination according to the clinical guidelines. Two doses will be given, in 3-week interval.

In these patients we will measure the specific antibody production. Blood sample 5 ml will be drawn before the first vaccine, before the second, and 3-4 weeks after the 2nd dose.

ELIGIBILITY:
Inclusion Criteria:

* Stem cell and and heart transplant patients who will receive pandemic H1N1 influenza vaccination according to the clinical guidelines.

Exclusion Criteria:

* Patients with unstable grafts.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Stem cell and and heart transplant patients who will receive pandemic H1N1 influenza vaccination according to the clinical guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-04 (Estimated); Study Completion 2010-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Engelhard, Principal Investigator — Hadassah
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel